CLINICAL TRIAL: NCT03796351
Title: A Randomized, Double-blind, Intra-Individual Controlled, Single-Center, Phase 1 Healthy Volunteer Study
Brief Title: Pharmacodynamic and Safety of MT10107(Botulinum Type A Neurotoxin) in Comparison to BOTOX®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: MT_PRT_EDB01
Record Dates: First submitted 2015-11-26; First posted 2019-01-08 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — coretox; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MT10107(botulinum toxin type A) (Experimental): Subjects will be administered a single equivalent dose of MT10107 by intramuscular injection to the EDB muscles of contralateral feet in five treatment group.
  Interventions: Drug: MT10107
- BOTOX® 50U(botulinum toxin type A) (Active Comparator): Subjects will be administered a single equivalent dose of BOTOX® 50U by intramuscular injection to the EDB muscles of contralateral feet in five treatment group.
  Interventions: Drug: Botox

INTERVENTIONS:
Drug: MT10107 — Subjects will be administered a single equivalent dose of MT10107 and Botox® by intramuscular injection to the EDB muscles of contralateral feet. Five cohorts of eligible subjects will be studied; Group A (2 U dose), Group B (5 U dose), Group C (10 U dose), Group D (20 U dose) and Group E (30 U dose).
  The foot in which each drug is to be administered (i.e. left or right) will be assigned in a randomized manner.
  Other Names: Coretox
  Arms: MT10107(botulinum toxin type A)
Drug: Botox — Subjects will be administered a single equivalent dose of MT10107 and Botox® by intramuscular injection to the EDB muscles of contralateral feet. Five cohorts of eligible subjects will be studied; Group A (2 U dose), Group B (5 U dose), Group C (10 U dose), Group D (20 U dose) and Group E (30 U dose).
  The foot in which each drug is to be administered (i.e. left or right) will be assigned in a randomized manner.
  Arms: BOTOX® 50U(botulinum toxin type A)

SUMMARY:
This study design is a randomized, double-blind, intra-individual controlled, single-center, phase 1 healthy volunteer study. Subjects who voluntarily signed the informed consent and are judged to be eligible for this study will be intramuscularly injected with the study drug or the comparator at a randomized unit(2U, 5U, 10U, 20U, 30U) in each site of the Extensor digirotum brevis. Thereafter, follow-up visits will be made 14 days, 30days, 60days, 90days and pharmacodynamic and safety assessments will be conducted for total 90days.

DETAILED DESCRIPTION:
This is a randomised, double-blind, intra-individual controlled, dose escalation study to assess the safety, tolerability and preliminary effectiveness of a single dose of MT10107 in comparison to Botox®50U (BOTOX® is a registered trademark owned by Allergan). This is the first-in-human study for MT10107, and will be performed in healthy volunteers.

Subjects will be administered a single equivalent dose of MT10107 and Botox®50U by intramuscular injection to the EDB muscles of contralateral feet. Five cohorts of eligible subjects will be studied; Group A (2 U dose), Group B (5 U dose), Group C (10 U dose), Group D (20 U dose) and Group E (30 U dose).

The foot in which each drug is to be administered (i.e. left or right) will be assigned in a randomized manner.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male adults aged between 20 and 65 years
2. Subjects with CMAP M-wave amplitude of the EDM muscle of ≥ 4.0 mV, CMAP M-wave amplitude of the AH muscle of ≥ 5.0 mV, and CMAP M-wave amplitude of the ADQ muscle of ≥ 5.0 mV.
3. Have no clinically significant medical conditions.
4. Able to provide written informed consent.
5. Able to attend all assessment visits.

Exclusion Criteria:

1. Subjects who have previously been treated in 3 month with botulinum toxin type A.
2. Subjects who had childhood botulism.
3. Subjects who have a pacemaker or other heart device.
4. Subjects who have had previous myotomy or denervation surgery in the muscle of interest (e.g., peripheral denervation and/or spinal cord stimulation).
5. Subjects with peripheral neuropathy and/or an accessary peroneal nerve.
6. Participation in any research study involving drug administration and/or significant blood loss.
7. Subjects with laboratory (haematology and biochemistry) or urinalysis results out of the normal range and considered to be of clinical significance by the investigator.
8. Subjects with a history of alcohol abuse and/or drug habituation.
9. Subjects who take regular medication.
10. Subjects with allergy or hypersensitivity to the investigational products or their components
11. Subjects who have been given any of the following drugs within previous 4 weeks at screening: Muscle relaxants, Benzodiazepines
12. Subjects who do not agree to use barrier method contraception (i.e. condoms) for the duration of the study.
13. Subjects who participate in regular physical activity/sport, which requires high load and intensity to the foot and cannot be stopped for the duration of the study.
14. Patients who are not eligible for this study at the discretion of the investigator

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
The percentage change in CMAP M-wave amplitude in EDB muscle compared with the individual mean baseline value. | 30 days after the injection
  percentage change of CMAP(Compound Muscle Action Potential) amplitude of the EDB(Extensor Digitorum Brevis) muscle from baseline

SECONDARY OUTCOMES:
The potential diffusion effect on the adjacent muscles (AH and ADQ) as measured by surface EMG. | 14, 30 and 90 days after the injection
  percentage change of CMAP(Compound Muscle Action Potential) amplitude of the adjacent muscles (AH and ADQ) from baseline
The percentage change in CMAP M-wave amplitude in EDB muscle compared with the individual mean baseline value. | 14 and 90 days after the injection
  percentage change of CMAP(Compound Muscle Action Potential) amplitude of the EDB(Extensor Digitorum Brevis) muscle from baseline

CONTACTS AND LOCATIONS:
Overall Officials: MyungEun Chung, Principal Investigator — Catholic University of Korea Saint Paul's Hospital
Locations (1):
- The Catholic University of Korea, St. Paul's Hospital, Seoul, South Korea